CLINICAL TRIAL: NCT04069559
Title: Developing Nursing Students Attitudes Towards Refugees Based on Contact Hypothesis: Study Protocol for a Randomized Controlled Trial
Brief Title: Migrant Health Promotion Program for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Tuba Demirel, Assistant Professor at Nursing Faculty, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019/101
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Refugees
Keywords: Refugees health; Contact hypothesis; Nursing students; Attitudes; Randomized controlled trial
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Who Masked: Outcomes Assessor
Masking Description: Blindness was done for data collectors and statistician. There were two group as intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention contain education and application about refugees health.
  Interventions: Other: To develop nursing students' attitudes towards refugees program which based on contact hypothesis.
- Control Group (No Intervention): Students of control group performed routine public health nursing practices.

INTERVENTIONS:
Other: To develop nursing students' attitudes towards refugees program which based on contact hypothesis. — In the first three weeks, education were given to the intervention group about refugees. Students watched a film on the theme of migration. After than the students contacted refugees in three different centers ( an immigrant health center, a school and a civil Society Organization) each of them for a total of nine weeks and two days a week.
  Arms: Intervention Group

SUMMARY:
The aim of the study is to determine effect of program about developing nursing students' attitudes towards refugees based on contact hypothesis on Xenophobia, Attitude towards Refugees and Intercultural Sensitivity.

DETAILED DESCRIPTION:
This Randomized Controlled Trials has been conducted with Bachelor's degree in nursing. Ninety students selected and randomly assigned to the intervention and control group as 45 students. Intervention group received a program about developing refugees health for 12 weeks. The content of this program consists of education and practices for refugees health.

Primary Outcome Measure: Xenophobia, Attitude towards Refugees and Intercultural Sensitivity Scale.

ELIGIBILITY:
Inclusion Criteria:

* The university students in the fourth year of nursing education

Exclusion Criteria:

* Refugees or immigrants students

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Xenophobia, | 12 weeks
  Xenophobia Scale: The scale consists of 11 items and a single factor structure. The lowest score that can be obtained from Likert type scale (6 options) is 14 and the highest score is 84; The higher the score, the higher the risk of xenophobia.
Attitude towards Refugees | 12 weeks
  Attitude towards Refugees Scale: The scale is a likert type (5 options) and has 5 sub-dimensions
Intercultural Sensitivity | 12 weeks
  Intercultural Sensitivity Scale: The scale consists of 24 items and is a five-point likert type. The lowest total score that can be obtained from the scale is 24 and the highest total score is 120. The increase in the total score obtained from the scale indicates that the level of cultural sensitivity increased.

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Akin, Professor, Study Director — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No